CLINICAL TRIAL: NCT02300701
Title: The Role of Anti-IgE (Omalizumab) in the Management of Severe Recalcitrant Paediatric Atopic Eczema
Brief Title: Role of Anti-IgE in Severe Childhood Eczema
Acronym: ADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADAPT
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Atopic Eczema; Atopic Dermatitis; Child
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xolair/Omalizumab (Experimental)
  Interventions: Drug: Xolair
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xolair — According to manufacturer's instructions
  Other Names: Omalizumab
  Arms: Xolair/Omalizumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of anti-IgE (Omalizumab/Xolair) in children with severe eczema.

DETAILED DESCRIPTION:
To address the value of anti-IgE in children with severe eczema.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 4-19 years
2. Severe eczema
3. Raised SpIgE or SPT to at least 1 food allergen or 1 aeroallergen AND/OR
4. Clinical impression that allergic exposures cause worsening eczema.
5. Total IgE level >300 kU/l
6. Clinically proven IgE-mediated allergic disease.
7. Written informed consent to participate.

Exclusion criteria:

1. Inability to comply with 2-4 weekly injections and clinic visits
2. Evidence of underlying immune compromise, autoimmune disease, immune complex mediated conditions.
3. Uncontrolled infection or unstable eczema.
4. Malignancy or a history of malignancy.
5. Pre-existing hepatic or renal impairment
6. Known cardiovascular or ischaemic cerebrovascular abnormality.
7. Other serious or uncontrolled systemic disease.
8. Pregnancy or lactation.
9. Known history of hypersensitivity or anaphylaxis to anti-IgE injections or its constituents.
10. Insufficient understanding of the trial assessments.
11. Participation in a CTIMP in the previous 60 days or (if known) 4 half-lives of the relevant medication, whichever is the greater.
12. Investigator feels that there is a good clinical reason why the child would be unsuitable.

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2014-12; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Improvement in atopic eczema | 24 weeks after treatment commences

CONTACTS AND LOCATIONS:
Overall Officials: S Chan, MBBS, MD, Principal Investigator — Guy's and St Thomas' Hospitals NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Chan S, Cornelius V, Cro S, Harper JI, Lack G. Treatment Effect of Omalizumab on Severe Pediatric Atopic Dermatitis: The ADAPT Randomized Clinical Trial. JAMA Pediatr. 2020 Jan 1;174(1):29-37. doi: 10.1001/jamapediatrics.2019.4476. PMID 31764962
- [Derived] Chan S, Cornelius V, Chen T, Radulovic S, Wan M, Jahan R, Lack G. Atopic Dermatitis Anti-IgE Paediatric Trial (ADAPT): the role of anti-IgE in severe paediatric eczema: study protocol for a randomised controlled trial. Trials. 2017 Mar 22;18(1):136. doi: 10.1186/s13063-017-1809-7. PMID 28330497